CLINICAL TRIAL: NCT03346798
Title: The Effect of Social Media on Eating Behaviours
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yale-NUS College (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YNC-CPST-03
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Food Photography; Non-Food Photography; No Phone Use
Keywords: External eating; Technology; Photography; Social media

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Photography (Experimental): On the first visit, participants will engage in food photography on their smart phones while eating. On the second visit, participants will not use their smart phones while eating.
  Interventions: Behavioral: Food Photography; Behavioral: No Phone Use
- Non-Food Photography (Experimental): On the first visit, participants will engage in non-food photography on their smart phones while eating. On the second visit, participants will not use their smart phones while eating.
  Interventions: Behavioral: Non-Food Photography; Behavioral: No Phone Use

INTERVENTIONS:
Behavioral: Food Photography — Participants will engage in food photography on their smart phones while eating
  Arms: Food Photography
Behavioral: Non-Food Photography — Participants will engage in non-food photography on their smart phones while eating
  Arms: Non-Food Photography
Behavioral: No Phone Use — Participants will not use their smart phones while eating

SUMMARY:
This project aims to explore how social media use, in particular food photography, influences eating behaviours. It will be approached through three methods - a correlational experience sampling method, an experimental experience sampling method, and an experimental laboratory method. This registration describes the experimental laboratory method.

DETAILED DESCRIPTION:
This project aims to explore how social media use, in particular food photography, influences eating behaviours.

The research question will be approached using a combination of methods. The first is the experience sampling method, where data is gathered from participants as they are going about their day-to-day lives. This method comprises two sub-sections - a correlational study, and an experimental study. The second approach is the experimental laboratory method, where participants will be randomly assigned to different conditions while given the opportunity to eat. This registration describes the experimental laboratory method.

Upon arrival at the lab, participants will first be required to fill in some online questionnaires (e.g. demographic information, mood rating scales). They will then be randomised to one of two conditions - to engage in food photography, or to engage in non-food photography - while eating some food and completing some rating scales. These photos will be taken with the intention of sharing on social media. Participants will then fill in some more online questionnaires, before leaving the lab. After the session, the amount of food consumed by the participants will be weighed.

As a control, all participants will be required to come back to the lab for a second visit one week later, where they will all complete the same eating and rating task, but without any phone use.

The expected outcome of the project is to collectively evaluate the data from the various methods to conclude how social media use, and in particular the act of food photography, influences the various aspects of eating behaviours.

ELIGIBILITY:
Inclusion Criteria:

- Instagram user

Exclusion Criteria:

* Symptoms / history of any medical or psychiatric conditions
* Allergies to food products
* History of eating disorders
* BMI: <18/ >28
* Excessive exercise (≥ 5 times a week of self-reported exercise)
* Currently on a special diet or deliberating restricting caloric intake
* Currently on a weight loss program

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-04-06 (Estimated); Study Completion 2018-04-06 (Estimated)

PRIMARY OUTCOMES:
Amount of food consumed | 12 minutes
  Weight of food after completing the lab session

SECONDARY OUTCOMES:
Enjoyment of food consumed | 12 minutes
  Self-reported rating between 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore